CLINICAL TRIAL: NCT00207103
Title: Phase I Dose Escalation Study to Determine the Safety, Pharmacokinetics and Pharmacodynamics of BMS-582664 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: MAD in Cancer Patients: Safety of BMS-582664 in Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA182-002
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2008-11-04 (Estimated); Status verified 2008-11

CONDITIONS: Tumors; Neoplasm Metastasis
Keywords: Advanced metastatic or solid tumors
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — brivanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental)
  Interventions: Drug: Brivanib
- 2 (Experimental)
  Interventions: Drug: Brivanib
- 3 (Experimental)
  Interventions: Drug: Brivanib
- 4 (Experimental)
  Interventions: Drug: Brivanib
- 5 (Experimental)
  Interventions: Drug: Brivanib
- 6 (Experimental)
  Interventions: Drug: Brivanab

INTERVENTIONS:
Drug: Brivanib — Tablets, Oral, 180 mg, once daily, until disease progression
  Other Names: BMS-582664
  Arms: 1
Drug: Brivanib — Tablets, Oral, 320 mg, once daily, until disease progression
  Other Names: BMS-582664
  Arms: 2
Drug: Brivanib — Tablets, Oral, 600 mg, once daily, until disease progression
  Other Names: BMS-582664
  Arms: 3
Drug: Brivanib — Tablets, Oral, 800 mg, once daily, until disease progression
  Other Names: BMS-582664
  Arms: 4
Drug: Brivanib — Tablets, Oral, 800 mg, once daily (5 days on, 2 days off), until disease progression
  Other Names: BMS-582664
  Arms: 5
Drug: Brivanab — Tablets, Oral, 1000 mg, once daily, until disease progression
  Other Names: BMS-582664
  Arms: 6

SUMMARY:
This is a Phase I dose escalation study to determine the safety, pharmacokinetics and pharmacodynamics of BMS-582664 in patients with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of progressive advanced or metastatic (tumor that has spread) solid tumors
* No tumor spread to the brain
* Feeling well other than cancer diagnosis (i.e. lab work, no infection, etc.)
* Available tumor tissue sample from prior surgery
* 4-6 weeks since prior therapy and recovered from prior therapy
* Men and women, ages 18 and above
* Women must not be pregnant or breastfeeding
* Diagnosis of advanced or metastatic (tumor that has spread) colorectal, hepatocellular (liver) or renal (kidney) cancer
* Measurable disease on scans (at least one)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2004-09; Primary Completion 2007-10 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety assessment | throughout the study
dose-limiting toxicity (DLT) | assessed for individual patients from C1D1 to C1D28 during the dose escalation portion of the protocol, until maximum tolerated dose is identified
determination of maximum tolerated dose (MTD) | during dose escalation portion of the protocol. Three to six subjects are treated at a specified dose level. If deemed safe dose escalation continues until the maximum tolerated dose is identified

SECONDARY OUTCOMES:
Efficacy based on duration of response and time to progression based on assessment | measured every 8 weeks throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- United States (3):
  - Premiere Oncology, Santa Monica, California
  - Indiana University Med Center, Indianapolis, Indiana
  - University Of Wisconsin Comprehensive Center, Madison, Wisconsin
- Canada (2):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Ottawa, Ontario
- Local Institution, Milan, Italy
- United Kingdom (2):
  - Local Institution, Middlesex, Greater London
  - Local Institution, Manchester, Greater Manchester